CLINICAL TRIAL: NCT01416272
Title: Twelve Month Clinical Evaluation of KeraSoft IC Soft Contact Lenses
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Study was terminated due to a business decision to cancel the entire project.
Sponsor: Bausch & Lomb Incorporated (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: ROC2-11-024
Record Dates: First submitted 2011-08-11; First posted 2011-08-15 (Estimated); Results first posted 2014-11-25 (Estimated); Last update posted 2014-11-25 (Estimated); Status verified 2014-11

CONDITIONS: Keratoconus
MeSH Terms: conditions — Keratoconus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- KeraSoft IC Soft Contact Lenses (Experimental): KeraSoft IC Soft Contact Lenses, with CIBA Clear Care solution provided for lens care
  Interventions: Device: KeraSoft IC Soft Contact Lenses

INTERVENTIONS:
Device: KeraSoft IC Soft Contact Lenses — Lenses will be worn between 8 and 16 hrs each day, for 12 months

SUMMARY:
The objective of this twelve month dispensing study is to evaluate the clinical performance, particularly comfort and vision, of KeraSoft IC Soft Contact Lenses.

ELIGIBILITY:
Inclusion Criteria:

* Have participated and completed a previous study (ROC2-10-078).
* Is Keratoconic

Exclusion Criteria:

* Has any systemic disease affecting ocular health.
* Is using any systemic or topical medications that will, in the Investigator's opinion, affect ocular physiology or lens performance.
* Is not correctable to 20/50 or better in each eye with contact lenses.
* Has greater than Grade 2 slit lamp exam findings.
* Has any atypical scar for a keratoconic or neovascularization within the central 4mm of the cornea. Subjects with minor peripheral corneal scarring that, in the Investigator's judgment, does not interfere with contact lens wear are eligible for this study.
* Has any neovascularization within the central 4mm of the cornea.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2011-04; Primary Completion 2012-12 (Actual); Study Completion 2013-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert Steffen, OD, MS, Study Director — Bausch & Lomb Incorporated
Locations (1):
- Bausch & Lomb Incorporated, Rochester, New York, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | KeraSoft IC Soft Contact Lenses
Started | 12
Completed | 8
Not Completed | 4
Not completed — Unacceptable distance visual acuity | 2
Not completed — Lost to Follow-up | 1
Not completed — Study related complaints | 1

BASELINE CHARACTERISTICS:
Arm/Group | KeraSoft IC Soft Contact Lenses
Number analyzed (Participants) | 12
Age, Continuous [Mean (Full Range); unit: years] | 48 [33 to 63]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 7

OUTCOME MEASURES:

1. Primary Outcome: Comfort
Description: Symptoms and complaints measured on an analog scale
Time Frame: 4 visits over 1 year
Population: DUE TO THE CANCELLATION OF THIS PROJECT, NO STATISTICAL OR CLINICALLY MEANINGFUL CONCLUSIONS RELATED TO THE STUDY ENDPOINTS WERE MADE.
Arm/Group | KeraSoft IC Soft Contact Lenses
Number analyzed (Participants) | 0

2. Secondary Outcome: Visual Acuity - Low Contrast
Description: Low contrast visual acuity measured with high ambient illumination (LCHI)
Time Frame: 4 visits over 1 year
Population: as for outcome 1
Arm/Group | KeraSoft IC Soft Contact Lenses
Number analyzed (Participants) | 0

3. Secondary Outcome: Visual Acuity - High Contrast
Description: High contrast visual acuity measured with high ambient illumination (HCHI)
Time Frame: 4 visits over 1 year
Population: as for outcome 1
Arm/Group | KeraSoft IC Soft Contact Lenses
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Arm/Group | KeraSoft IC Soft Contact Lenses
Serious Adverse Events (participants affected / at risk) | 0/12
Other Adverse Events (participants affected / at risk) | 0/12

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes